CLINICAL TRIAL: NCT05465174
Title: Tovorafenib for the Treatment of Newly Diagnosed or Recurrent Craniopharyngioma in Children and Young Adults
Brief Title: Tovorafenib for Treatment of Craniopharyngioma in Children and Young Adults
Acronym: PNOC029
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sabine Mueller, MD, PhD (Other)
Collaborators: Day One Biopharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Sabine Mueller, MD, PhD, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 210828; NCI-2022-05356 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2022-07-15; First posted 2022-07-19 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Craniopharyngioma, Child; Craniopharyngioma; Recurrent Craniopharyngioma
Keywords: Neoadjuvant therapy
MeSH Terms: conditions — Craniopharyngioma | interventions — tovorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: Neoadjuvant Tovorafenib (Experimental): Participants with newly diagnosed craniopharyngioma will receive one (1) dose of Tovorafenib within 7 days +/- 2 days prior to planned biopsy or resection. At completion of biopsy or resection, participants having undergone biopsy only or sub-total (STR) or near-total resection (NTR) will continue on maintenance monotherapy of Tovorafenib given once weekly at the respected recommended phase 2 dose (RP2D). Participants having undergone a gross total resection (GTR) will enter into follow-up only and will be part of the exploratory cohort.
  Interventions: Drug: Tovorafenib
- Group 2, Arm A: Neoadjuvant Tovorafenib (Experimental): Participants with recurrent craniopharyngioma will receive one (1) dose of Tovorafenib within 7 days +/- 2 days prior to planned biopsy or resection. At completion of biopsy or resection, participants having undergone biopsy only or STR or NTR will continue on maintenance monotherapy of Tovorafenib given once weekly at the respected RP2D.
  Interventions: Drug: Tovorafenib
- Group 2, Arm B: Non-biopsy/resection participants (Experimental): Non-biopsy/resection participants with recurrent disease will receive monotherapy of Tovorafenib given once weekly at the respected RP2D.
  Interventions: Drug: Tovorafenib

INTERVENTIONS:
Drug: Tovorafenib — Given orally
  Other Names: DAY101; TAK580; AMG-2112819; BSK1369

SUMMARY:
The current study assesses the tolerability and efficacy of monotherapy with pan-RAF-kinase (Tovorafenib) inhibition for the treatment of children and young adults with craniopharyngioma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine progression free survival and maintenance of quality of life at 12 months as based on physical function and compared to historical controls.

SECONDARY OBJECTIVES:

I. To identify proportion of participants with visual deficits at 1-year, 2-year, and 3-year follow-up.

II. To identify proportion of participants with neuroendocrine deficits at 1-year, 2-year, and 3-year follow-up.

EXPLORATORY OBJECTIVES:

I. To assess Quality of Life (QOL) and cognitive measures in children and young adults with newly diagnosed or recurrent craniopharyngioma.

II. To perform Immunohistochemistry (IHC)/Multiplexed ion beam imaging on pre-and post-treatment tumor tissue (as available), including at time of progression, to assess for patterns of protein density and spatial relationship in intact tumor tissue and elucidate changes in tumor tissue over the course of therapy and disease evolution.

III. To perform single-cell (scRNA) RNA sequencing on pre- and post-treatment tumor tissue (as available), including at time of progression, to identify and characterize distinct cell subsets that make up the components of craniopharyngioma and elucidate changes in cell subsets over the course of therapy and disease evolution.

IV. To perform proteomic analysis on pre- and post-treatment tumor tissue, including at time of progression, to characterize distinct proteins and transcriptome pathways that are active in different tumor compartments and elucidate changes in proteomic profiles over the course of therapy and disease evolution.

V. To perform ELISA array/multiplex analysis on pre- and post-treatment cyst fluid, including at time of progression, to characterize distinct cytokine profiles and elucidate changes in cytokine profile over the course of therapy and disease evolution.

VI. Microbiome and flow cytometry studies in the context of imaging and clinical outcomes using descriptive statistics.

VII. To assess patient and/or proxy satisfaction with study participation via patient-reported outcome (PRO) measures.

VIII. To assess patient and/or proxy satisfaction with study participation via patient-reported outcome (PRO) measures in the context of race ethnicity and other health related social risks.

IX. To assess on therapy toxicity in the context of race, ethnicity and other health related social risks.

TREATMENT GROUPS:

Participants will be divided into 2 cohorts: newly diagnosed or recurrent craniopharyngioma, both planned for standard of care biopsy/resection. All newly diagnosed participants or recurrent craniopharyngioma without histologic diagnosis will be enrolled on a screening consent for central imaging review to ensure imaging supports diagnosis of craniopharyngioma before enrollment onto the treatment protocol. After enrollment onto treatment protocol, each patient in each arm will receive one dose of tovorafenib prior to planned biopsy or resection. Participants with measurable disease will then continue on maintenance therapy. Participants who have a gross total resection (GTR) will enter into the follow-up only phase.

ELIGIBILITY:
Inclusion Criteria:

Newly Diagnosed Participants:

* Newly diagnosed craniopharyngioma, as based on imaging characteristics and central radiology review. Participants will initially be screened within confines of a screening consent and only those participants with findings consistent with craniopharyngioma and without findings suggesting an indeterminate lesion or lesion of an alternative diagnosis (including abnormal tumor markers found in blood or cerebral spinal fluid (CSF), if completed as part of standard of care (SOC) work-up or if lesion concerning for alternate diagnosis) will move ahead with enrollment on the treatment protocol. Additionally, for participants that have undergone initial biopsy to confirm diagnosis, are within 6 weeks of radiographic diagnosis, and are planned to undergo follow up second surgery for additional tumor resection as per standard of care recommendations, these participants will also be considered eligible.
* Participants must be surgical candidates for biopsy or resection and planned for standard of care biopsy or resection.

Recurrent Participants:

* Recurrent craniopharyngioma, as based on histologic confirmation at time of initial diagnosis (participants with Adamantinomatous craniopharyngioma (ACP) will only be eligible for the recurrent arm).
* Recurrent craniopharyngioma without prior histologic confirmation will initially be screened within confines of a screening consent and only those participants with findings consistent with craniopharyngioma and without findings suggesting an indeterminate lesion or lesion of an alternative diagnosis (including abnormal tumor markers found in blood or CSF, if completed as part of SOC work-up or if lesion concerning for alternate diagnosis) will move ahead with enrollment on the treatment protocol.
* Participants should be surgical candidates for biopsy or resection. If participants are not surgical candidates, but have available archival tumor tissue, they will be enrolled into the exploratory cohort.
* Participants must be willing to provide archival tissue, a minimum of 10-20 paraffin embedded unstained slides OR 1 block with tumor content of 40% or greater is required. Participants who do not meet this criteria may be discussed on a case-by-case basis with the Study Chair(s).
* Participants can have been previously treated with surgical resection alone, cyst drainage and biopsy alone, radiation therapy, other systemic therapies, or any combination thereof.
* Prior Therapy:

  * Had their last dose of myelosuppressive chemotherapy >= 21 days prior to study registration (>=42 days if nitrosourea therapy).
  * Had their last dose of hematopoietic growth factor >=14 days (long-acting growth factor) or >=7 days (short-acting growth factor) prior to study registration, or beyond the time during which adverse events (AEs) are known to occur.
  * Had their last dose of biologic (anti-neoplastic agent) >=7 days prior to study registration, or beyond the time during which AEs are known to occur.
  * Had their last dose of monoclonal antibodies >=21 days prior to study registration.

Radiation:

* Had their last fraction of local irradiation to primary tumor >=12 weeks prior to registration; investigators are reminded to review potentially eligible cases to avoid confusion with pseudo-progression.
* At least 14 days after local palliative radiation (small-port).

All Participants:

* Age 1 to 39 years.
* Participants continuing on maintenance therapy after standard of care biopsy/resection must have measurable disease, as defined as lesions that can be accurately measured in two dimensions (longest diameter to be recorded) with a minimum size of no less than double the slice thickness. Previously irradiated lesions are considered non-measurable except in cases of documented progression of the lesion since the completion of radiation therapy. Participants without measurable disease may continue on study and will be followed for study endpoints, but will not be included as part of target accrual.
* Performance Score: Karnofsky >= 50 for participants > 16 years of age and Lansky >= 50 for participants <= 16 years of age. Participants who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Corticosteroids: Participants who are receiving dexamethasone must be on a stable or decreasing dose for at least 1 week prior to registration. The participant steroid dose should be no more than a steroid-equivalent of dexamethasone 0.1 mg/kg/day (or maximum 4mg/day; whichever is the lower dose) at time of enrollment. Participants that have been stable on physiologic hormone replacement for hypopituitarism are allowed.
* Organ Function Requirements:

  * Adequate Bone Marrow Function defined as:

    * Peripheral absolute neutrophil count (ANC) >=1000/mm3.
    * Platelet count >= 100,000/mm3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment).
  * Adequate Renal Function defined as-

    ---A serum creatinine < 1.5 Upper Limit normal (ULN) based on age and gender.
  * Adequate Liver Function defined as-

    * Bilirubin (sum of conjugated + unconjugated) <= 1.5 x upper limit of normal (ULN) for age (except in participants with documented Gilbert syndrome).
    * Serum glutamic-pyruvic transaminase (SGPT)((alanine aminotransferase (ALT)) <= 3 x ULN.
    * Serum albumin >=2 g/dL (20g/L).
  * Adequate Neurologic Function defined as participants with seizure disorder may be enrolled if well controlled. Participants on non-enzyme inducing anticonvulsants may be excluded pending interaction(s) with study drug.
  * Adequate Pulmonary Function defined as no evidence of dyspnea at rest, no exercise intolerance due to pulmonary insufficiency, and a pulse oximetry of > 92% while breathing room air.
  * prothrombin time (PT) /partial thromboplastin time (PTT)/International Normalized Ratio (INR) within institutional normal limits or deemed appropriate for surgical intervention by the treating team for patients undergoing surgery biopsy/resection
* The effects of Tovorafenib on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (non-hormonal contraception; barrier method of birth control; abstinence - note, tovorafenib can make hormonal contraceptives ineffective) prior to study entry, for the duration of study participation and 28 days after completion of Tovorafenib administration, whichever is later. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* A legal parent/guardian or participants must be able to understand, and willing to sign, a written informed consent and assent document, as appropriate.
* Ability to complete the PedsQL Core Module. Patients must enroll on PNOC COMP if PNOC COMP is open to accrual at the enrolling institution.

Exclusion Criteria:

Newly Diagnosed Participants:

- Participants should not have undergone any previous tumor-directed therapy.

Recurrent Participants:

* Participants who have had chemotherapy or radiotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from acute adverse events due to agents administered more than 4 weeks earlier.
* Participants must be at least 1 week since the completion of therapy with a biologic or small molecule agent. For any agent with known adverse events that can occur beyond 1 week after administration, the period prior to enrollment must be beyond the time during which adverse events are known to occur. Such participants should also be discussed with study chairs.
* Participants should not have previously received any RAS-pathway, but have not received Tovorafenib will be eligible.

All Participants:

* Rapidly progressive symptoms that require urgent surgery or radiation therapy, which would prevent central review and or preclude participation with tumor-directed medical management alone.
* Uncontrolled symptoms of neuroendocrine dysfunction such as diabetes insipidus, hypothyroidism, panhypopituitarism (participants can be on supplemental medications for hormonal repletion; however, should be on controlled doses for at least 2 weeks prior to enrollment).
* Clinically significant active cardiovascular disease, or history of myocardial infarction, or deep vein thrombosis/pulmonary embolism within 6 months prior to registration, ongoing cardiomyopathy, or current prolonged QT interval corrected for heart rate by Fridericia's formula (QTcF) interval > 440 ms based on triplicate ECG average.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Tovorafenib or other agents used in study.
* Nausea and vomiting >= Grade 2, malabsorption requiring supplementation, or significant bowel or stomach resection that would preclude adequate absorption.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection.
* Participants who are receiving any other investigational agents.
* Women of childbearing potential must not be pregnant or breast-feeding.
* Current treatment with a strong cytochrome P4502C8(CYP2C8) inhibitor or inducer other than those allowed per Section 5.6.1. Medications that are substrates of CYP2C8 are allowed but should be used with caution.
* Participants with inability to return for follow-up visits or obtain follow-up studies required to assess toxicity to therapy.

Ages: 1 Year to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 57 (Estimated)
Dates: Start 2022-09-12 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival rate (PFS) | Up to 12 months
  Progression-free survival is defined as the time of documented response until disease progression as defined by Response assessment in neuro-oncology criteria (RANO) criteria. PFS will be reported by overall group at 12 months.
Changes in scores on the Physical functioning subscale of the Pediatric Quality of Life Inventory (PedsQL) over time | Up to 12 months
  Scores over time from the PedsQL 4.0 Generic Core physical function domain rating form, which have multidimensional child self-report and parent proxy report scales to assess health-related quality of life (QOL) in children, adolescents, and young adults ages 2 - 25 years will be reported. Physical functioning, is the sub-scale of interest for this protocol. Items on the physical functioning sub-scale are scored on a 5-point Likert scale with raw scores ranging from 0- 4. Items are reversed scored and linearly transformed to a 0-100 scale. If more than 50% of the items in the scale are missing, the Scale Scores should not be computed. Higher scores indicate a higher level of physical functioning

SECONDARY OUTCOMES:
Proportion of participants with visual deficits over time | Up to 5 years
  Teller acuity testing using Teller Acuity Cards® (TAC) II will be performed on every time participants undergo a radiographic disease assessment. Visual acuity (VA) testing will be performed in each eye separately at a distance of 55 centimeters in all participants. The tester will use the "two down, one up" protocol to achieve the best VA score. Acuity will be reported in logarithm of the minimum angle of resolution (logMAR). Visual field testing will be performed by confrontation and reported as the number of quadrants (0, 1, 2, 3, or 4) with visual field deficits. Optic discs will be assessed for the presence or absence of pallor and edema.The proportion of participants with recorded visual deficits over time based on these assessments will be reported.
Proportion of participants with neuroendocrine deficits | Up to 5 years
  The proportion of participants with presence of new neuroendocrine deficits defined as hypothalamic obesity, diabetes insipidus, growth hormone deficiency, adrenal insufficiency from baseline will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Mueller, MD, PhD, MAS, Principal Investigator — University of California, San Francisco; Cassie Kline, MD, Study Chair — Children's Hospital of Philadelphia
Locations (17):
- United States (15):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Rady Children's Hospital/University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - University of Florida, Gainesville, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana
  - John Hopkins University, Baltimore, Maryland
  - Dana-Farber/Boston Children's Harvard Medical School, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Children's Minnesota, Minneapolis, Minnesota
  - St. Louis Children's Hospital Washington University, St Louis, Missouri
  - NYU Langone Health, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah
- Australia (2):
  - Children's Cancer Centre, Monash Children's Hospital, Clayton, VIC 3168
  - Perth Children's Hospital, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data after de-identification may be shared with other researchers.
Supporting Information: Study Protocol